CLINICAL TRIAL: NCT06357416
Title: The Man Van Project: An Evaluation of the Effectiveness of a Mobile Outreach Screening Clinic Model for Earlier Detection of Prostate Cancer and Other Male Cancers
Brief Title: The Man Van Project
Acronym: MV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: RM Partners West London Cancer Alliance (Unknown); Institute of Cancer Research, United Kingdom (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCR5573
Record Dates: First submitted 2024-03-22; First posted 2024-04-10 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer; Urologic Cancer; Urologic Diseases; Bladder Cancer; Diabetes; Hypertension; Mental Health Issue; Alcoholism; Smoking; Renal Cancer; Testis Cancer
Keywords: mobile health; targeted screening
MeSH Terms: conditions — Prostatic Neoplasms; Urologic Neoplasms; Urologic Diseases; Urinary Bladder Neoplasms; Diabetes Mellitus; Hypertension; Alcoholism; Smoking; Kidney Neoplasms; Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Main Group (MV-Eco) Sub-study (Other): Patients seen in the Man Van, including those consenting to long-term follow-up of data.
  Interventions: Other: Main Man Van Group Sub-study (MV-Eco); Other: Man Van patients
- Point of care testing (MV-POCT) Sub-study (Other): Patients consenting to a point of care blood test for either a PSA and/or HbA1c
  Interventions: Device: MV-POCT Sub-study; Other: Man Van patients
- Qualitative questionnaire (MV-QualQ) Sub-study (Other): Patients consenting to participate in a qualitative study about their experience of the Man Van.
  Interventions: Other: MV-QualQ Sub-study; Other: Man Van patients
- Polygenic risk scores (MV-PRS) Sub-study (Other): Patients consenting for a polygenic risk score test.
  Interventions: Diagnostic Test: MV-PRS Sub-study; Other: Man Van patients
- DNA Collection (MV-DNA) and Urinary Circulating Tumour DNA collection (MV-UctDNA) Sub-studies (Other): Patients consenting to collection of DNA and/or urine for as yet undetermined future ethically-approved research.
  Interventions: Other: MV-DNA and MV-UctDNA Sub-study; Other: Man Van patients
- Man Van patients (Other): All patients seen within Man Van
  Interventions: Other: Man Van patients
- Stakeholder service interviews (MV-SSI) Sub-Study (Other): Semi-structured interviews with people involved in the running of the project or those who may help in recruiting patients. This may include but not be limited to: GPs, community leaders (e.g. church pastors), charity leaders, staff involved in delivery (nurses, co-ordinators), men who did not attend the service and relatives of men.
  Interventions: Other: MV-SSI Sub-study
- Target product profile (MV-TPP) Sub-Study (Other): We will develop an equity-focused Target Product Profile (TPP) that can provide a summary of the requirements for an optimal yet realistic profile of biomarker tests designed to work in mobile testing clinics, such as the Man Van.
  Interventions: Other: Man Van patients; Other: MV-TPP Sub-study

INTERVENTIONS:
Device: MV-POCT Sub-study — Point of care blood testing
  Arms: Point of care testing (MV-POCT) Sub-study
Other: Main Man Van Group Sub-study (MV-Eco) — Consent for long-term follow-up of patients
  Arms: Main Group (MV-Eco) Sub-study
Other: MV-QualQ Sub-study — Qualitative questionnaire and interview sub-study
  Arms: Qualitative questionnaire (MV-QualQ) Sub-study
Diagnostic Test: MV-PRS Sub-study — Patients consenting to polygenic risk score testing
  Arms: Polygenic risk scores (MV-PRS) Sub-study
Other: MV-DNA and MV-UctDNA Sub-study — Patients consenting to collection of DNA and urine for further study.
  Arms: DNA Collection (MV-DNA) and Urinary Circulating Tumour DNA collection (MV-UctDNA) Sub-studies
Other: Man Van patients — All patients seen in Man Van
  Arms: DNA Collection (MV-DNA) and Urinary Circulating Tumour DNA collection (MV-UctDNA) Sub-studies; Main Group (MV-Eco) Sub-study; Man Van patients; Point of care testing (MV-POCT) Sub-study; Polygenic risk scores (MV-PRS) Sub-study; Qualitative questionnaire (MV-QualQ) Sub-study; Target product profile (MV-TPP) Sub-Study
Other: MV-SSI Sub-study — Semi-structured interviews will be conducted with stakeholders involved in the running of or recruitment to the project.
  Arms: Stakeholder service interviews (MV-SSI) Sub-Study
Other: MV-TPP Sub-study — Multi-stage qualitative study comprising of interviews and participatory design focus group workshops.
  Arms: Target product profile (MV-TPP) Sub-Study

SUMMARY:
National Health Service (NHS) England has commissioned The Royal Marsden Hospital NHS Foundation Trust to run a novel mobile clinical outreach service called 'Man Van' with the aim of enabling male patients' easy access to care at the site of their work and in their communities. The initial focus of this new standard of care clinic is to access workplaces with large manual workforces where large scale working from home is not possible. These will include logistics firms and bus companies. These companies employ large numbers of black and minority ethnic men who also have poorer outcomes with a range of other diseases, including Coronavirus disease (COVID)-19. The novel clinical service will collaborate with Unite (and other unions) as well as employers in order to reach our target groups effectively. There is also the opportunity to target higher risk groups e.g. Afro Caribbean communities whose rates of prostate cancer are 1 in 41 as well as occupational higher risk categories. The Man Van has the potential to swing the balance of evidence in favour of Prostate-Specific Antigen (PSA) screening, with a targeted screening program directed at high-risk groups including ethnic minorities and manual workers. Reasons for poorer outcomes amongst these groups are multi-factorial and complex. Levels of education are often a factor which can impact the understanding of the disease and how to seek assistance. Distrust of medical organisations has also been cited as a factor.

The aim of the Man Van mobile outreach service is to enable men access to a specific men's health service - focusing on general health and wellbeing (including BMI assessment, blood pressure, blood sugar/diabetes checks etc) and a prostate check for those who raise concerns. This will include a PSA test where relevant. This will be the core data gathered from the project.

Patients will receive PSA results in the 'Man Van' by a clinical nurse specialist with patients with raised PSA levels being referred into the standard rapid referral cancer pathways. Similar considerations will apply to men with haematuria detected on dip stick testing or who present with a testicular mass or penile lesion (both rare but important).

The clinical data generated from each routine health screening appointment will be analysed to determine the effectiveness of the Man Van mobile outreach model in identifying prostate and other male cancers and other co-morbidities much earlier than if patients had waited to present to their General Practitioner (GP) or other healthcare provider.

Patients who receive an early diagnosis of clinically significant prostate cancer will have access to early curative treatments, which are typically less invasive and shorter in timescales. Similar interventions have shown large scale success in particular with breast and cervical cancer.

The NHS sees many patients accessing cancer care at a late stage. Reducing this trend is a key objective of the NHS Long Term Plan. The COVID-19 pandemic has further exacerbated health inequalities and mobile clinics can potentially be a model for alleviating this. To enable patients access to medical treatment earlier there is a need to make the 'seeking advice on men's health and prostate issues' less daunting, more normal and easily accessible. The 'Man Van' has the ability to do just that and it is anticipated that the findings of this research, using the data generated from each patient's routine health screening, will demonstrate that a mobile outreach model is more effective in identifying cancers at an earlier stage than 'traditional' diagnostic pathways.

We also hope to evaluate the Man Van with a qualitative study looking at the patient perspectives from those who utilise the Man Van.

The reasons for high risk in prostate cancer are heavily linked to genetics. This is an issue as there is less recruitment of high risk groups to studies. We hope to gather genetic data from a higher proportion of genetically susceptible men via the Man Van, which can be used in future to further genetic knowledge of prostate cancer.

DETAILED DESCRIPTION:
Background

Early intervention is potentially lifesaving for a range of conditions. A key cause of death from cancer and other causes is late presentation and there are key barriers to early access such as low education levels, difficult access to primary care (for example due to anti-social working hours) as well as lack of knowledge of relevant symptoms that might trigger referral and investigation. The Man Van project seeks to address some of these reasons for late presentation and started with an initial focus on prostate cancer. The project has now broadened to include a range of conditions that are major causes of mortality and morbidity in men such as heart and liver disease, other urological cancers (penile, testicular, bladder, kidney). The Man Van clinics will be focused on populations at risk of delayed presentation to healthcare systems such as men in manual or low skill jobs and workplaces with high numbers of black and ethnic minority employees.

Prostate cancer is the most common cancer in men in the United Kingdom (UK), with over 50,000 new cases diagnosed and 15,000 lives lost to prostate cancer in the UK each year 1. This is of particular concern for black African and African Caribbean men who carry a 1 in 4 risk of developing prostate cancer, and for men with a family history of the disease. Another challenge is that, typically, men tend to approach their GP for men's health issues when symptoms are severe. Around 20-25% of men with prostate cancer still present to A&E with retention. At this late-stage treatment is less likely to be successful and certainly will carry more morbidity for the patient and cost for the health care system. The recent COVID-19 pandemic has further exacerbated this issue with routine referrals to cancer diagnostics clinics dropping by around a third (in house data, Royal Marsden Hospital), suggesting a growing reservoir of un-diagnosed cancer in the community.

Till date there is no consensus on the modality of prostate cancer screening, but most studies have focussed on PSA as a screening tool, with MRI scanning and biopsies as adjuncts to this. PSA itself has a controversial history in screening for prostate cancer with studies showing differing results. A key issue in using PSA as a screening tool comes from the definition of what a 'normal' PSA is. PSA increases with age and with benign growth of the prostate but can also be elevated in urinary tract infections or prostatic inflammation. Oesterling's age specific PSA ranges from 1993 are still in use today. Prostate cancer is of course another cause of PSA elevation. Having a higher PSA threshold for investigation increases the positive predictive value for detecting prostate cancer but lowers the negative predictive value, and the reverse is true as well. A study by Gerstenbluth documented a positive predictive value of 98.5% for PSA in detecting prostate cancer with a PSA of 50ng/ml or above.

The evidence for screening is also controversial resulting in differing guidance around the world. The Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial from the USA looked at systematic vs opportunistic screening in over 76000 men. Using a PSA threshold of over 4 and 7-10 years of follow-up no significant difference in mortality from prostate cancer was found between the screened and non-screened arms. However, the study had high rates of contamination between the two groups with an estimated 74% of the control group subject to at least one routine PSA test during the trial (95% in the intervention arm) and around 50% of men in the control group tested each year.

The European Randomized Study of Screening for Prostate Cancer (ERSPC) has been studying 186,000 men aged 55 to 69 in Europe since 1992. Now in its 16th year of follow-up6 results show a 20% reduction in cancer specific survival, and the numbers needed to treat was now below that which is observed in breast cancer strengthening the argument for some form of screening. A total of seven studies in different regions of Europe were included, with each study utilising different screening criteria and treatment protocols, interval timing, and PSA cut-offs (between 3 and 4), again muddying the waters. As a result of this conflicting evidence the National Institute of Clinical Excellence (NICE) guidelines suggest a risk stratified approach along with patient counselling. The guidelines recommend giving a PSA test to any man over the age of 50 years who requests it as well as offering it to men with lower urinary tract symptoms, haematuria, erectile dysfunction or symptoms that may suggest advanced prostate cancer such as unexplained bone pain or weight loss. However, routine systematic screening is not recommended.

Rationale

The rationale behind the introduction of the Man Van mobile outreach service is to increase patient access and support to cancer investigation pathways. This is particularly important in patient groups from lower socio-economic and high risk groups where delay in early intervention can result in delayed presentation and adverse health outcomes. We hope to demonstrate the feasibility and applicability of such a service to improve patient outcomes and hope to gather important qualitative and DNA based data for further research.

This research project will analyse the clinical data obtained from each patient's routine health screening and long-term follow-up data from NHS Digital and other healthcare providers, to make a full assessment of how effective the Man Van mobile outreach model is in diagnosing prostate and other male cancers by making a comparison with the current detection rates from diagnoses made under the traditional screening and diagnosis pathway. It is anticipated that the results of this study will provide further evidence for the commissioning of targeted outreach programmes for early detection of prostate and other male cancers.

Point of care testing (MV-POCT)

Point of care blood testing is a feature of the van that will allow instant results to be given to patients, preventing the need for follow-up appointments and speeding up diagnoses. Both PSA and HbA1c tests are currently carried out on the van using formal laboratory blood tests which are then sent via courier to the Royal Marsden biochemical laboratory.

As well as a formal laboratory validation process which is required before any point of care machine can be used (which is not part of the research protocol) we will determine what effect the difference between laboratory and point of care testing may have on the decision making process for patients.

The clinical decision making from PSA testing will be whether an onwards referral for prostate cancer investigation is recommended by the clinical team. For HbA1c it will be whether a primary care referral for diabetic management is recommended by the clinical team. The laboratory value will be taken as the 'true' value in this instance as all final clinical decision making based on this.

Qualitative questionnaire (MV-QualQ)

As the Man Van provides a new clinical model for assessing patients, the patients' perspective on the model, and comparisons to existing clinical services is important. Going into more detail than a service evaluation questionnaire, a qualitative study has been developed to better understand how patients feel about and react to the service. A qualitative questionnaire has been developed following discussion group input via a modified Delphi process.

The Delphi method is a commonly used method for achieving a consensus of opinion of real world knowledge from experts in the field. It was developed by Dalkey and Helmer at the Rand Corporation in the 1950s and is aimed at problem-solving, idea-generation, or determining priorities.

The complexity of issues that prevent men from seeking or finding healthcare and our lack of understanding is the key driver for this study. This is particularly relevant for men from ethnic minorities and lower socio-economic groups. Understanding the barriers and facilitators to healthcare access may provide further support of the Man Van project and may help develop further research themes aimed at increasing healthcare access.

In-depth qualitative patient interviews will be carried out on at least 5 patients to further delineate themes which arise from the questionnaires. With permission interviews will be recorded and transcribed to aid thematic analysis.

Health Economic Analysis (MV-Eco)

A key element of the Man Van project is its long-term use as a novel method of targeted screening and improving health care outcomes. Like all NHS funded services a cost-benefit analysis is integral to supporting the case for this project into the future. Health economic arguments form key parts of discussion for NICE and NHS England commissioning groups.

The health economic arguments for prostate cancer screening remain unclear as they do for various diseases, however a combined approach that targets high risk patients and assess for prostate cancer, bladder/renal cancer, diabetes, hypertension and other diseases assessed for in the Man Van may make for a stronger economic argument.

Polygenic risk scores (MV-PRS)

Prostate cancer is the commonest cancer in men in the Western world, with over 40,000 new cases per annum. However, its aetiology remains very poorly understood. The substantial variation in incidence rates worldwide suggests that lifestyle risk factors are important however, no definite lifestyle risk factors have been identified till date.

Family history has been identified as a significant risk factor for prostate cancer, as it is in many other cancers and diseases. Although this is likely due to inherited genetic pre-disposition, causation is yet to be fully established.

Although gene mutations have been discovered as being causative factors for many diseases PRS allow for the amalgamation of greater variants in order to explain a larger proportion of diseases rather than single low penetrance variants. PRS has the potential to enhance risk susceptibility to a greater proportion of the population and offer new avenues in patient screening and disease prevention.

The clinical application of PRS is subject of intense debate and ongoing research. We hope to add to this area of ongoing study, in particular with the combination of offering lifestyle modification advice in the context of PRS. PRS scores will be generated from saliva samples of DNA. As is common with many studies the under recruitment and under representation of ethnic minority patients remains an issue, resulting in less representative polygenic risk scores for patients of non-white ethnicities. We hope to address this via the Man Van by recruiting higher proportions of other ethnicities.

DNA Collection (MV-DNA)

Genetic studies have become a key part of cancer research, both for early diagnosis and prognostic reasons. A key issue for studies is trial recruitment, with significant issues in the recruitment of ethnic minorities to trials, which is particularly relevant when a disease may affect a particular ethnicity more (for example prostate cancer in Black men). DNA collection with either blood or saliva samples can help to build a database which can be used for further genetic studies.

Urinary Circulating Tumour DNA collection (MV-UctDNA)

Despite much research into the development of novel urinary biomarkers for bladder cancer, the mainstay of diagnosis remains invasive with a flexible (or rigid) cystoscopy. Even cystoscopy is only carried out after a red flag symptom triggers a referral (haematuria or recurrent infections). Several tests exist but none has replaced cystoscopy as the gold standard either for diagnosis of new bladder cancer or disease recurrence. Circulating tumour DNA (ctDNA) from urine has potential as a new avenue of development of diagnostic tests for bladder cancer and also prostate cancer.

ELIGIBILITY:
Patients are eligible to be included in the research study if they are eligible to access the Man Van mobile outreach clinic, which is a novel clinical service delivered by The Royal Marsden Hospital NHS Foundation Trust. The inclusion and exclusion criteria have been designed to be as broad as possible, in order to include data from as many patients using the Man Van clinical service as possible.

As the primary purpose of the Man Van mobile outreach clinic is to screen for prostate, testicular, penile and other cancers that affect men, only men are eligible to be reviewed in the mobile outreach clinic hence only males will be recruited into this study.

Inclusion criteria for the Main Study

1. Participating in the linked Man Van mobile outreach clinic
2. Age ≥45 years
3. Male

   (The initial pilot study had a age criteria of ≥18 years, but this was amended).

   MV-POCT

   Inclusion Criteria: Any patient having a PSA and/or an HbA1c test as part of a Man Van work up, or via the our rapid diagnostics clinic.

   MV-QualQ

   Inclusion Criteria: Any patient attending the Man Van for an assessment.

   MV-Eco

   Inclusion Criteria: Any patient attending the Man Van for an assessment.

   MV-PRS

   Inclusion Criteria: Any patient attending the Man Van for an assessment and able to provide saliva samples.

   MV-DNA

   Inclusion Criteria: Any patient attending the Man Van for an assessment, and able to provide blood/saliva samples.

   MV MV-UctDNA

   Inclusion Criteria: Any patient attending the Man Van for an assessment, and able to provide urine samples.

   MV-SSI

   Inclusion criteria:
   * Aged > 18 and over (on date of invitation to participate)
   * Works for healthcare organisation, other stakeholder or professional or potential man van patient who was not seen or relative of a Man Van patient/potential patient

   Exclusion criteria:
   * Man van patient who has attended appointment

   MV-TPP

   Inclusion criteria:

   Healthcare Professionals
   * Aged > 18 and over (on date of invitation to participate)
   * Speaks English
   * Works within the UK
   * Profession: GPs, Practice Staff (Nurses, Physician Assistants and Associates
   * Healthcare assistants)
   * Experienced in adopting new tests and guidelines into practice.
   * Experienced in detecting, managing, and referring symptoms and asymptomatic patients with symptoms of prostate, pancreatic, GI cancer and/or are at an increased risk of developing these cancers.

   Patients
   * Aged > 18 and over (on date of invitation to participate)
   * Speaks English
   * Lives in the UK
   * Patients with direct and in-direct experience with prostate, pancreatic, GI cancers.
   * Patients at an increased risk of developing prostate, pancreatic, GI cancer in accordance with known risk factors, which includes age, smoking, being overweight or obese, family history and genetic factors, pancreatitis, and diabetes.

   Other key stakeholders/professionals

   • Aged > 18 and over (on date of invitation to participate)

   • Speak English
   * Works within the UK
   * Professions: medical devices and biomedical researchers, scientists, representatives for major regulatory and funding bodies
   * Knowledgeable of Early Detection initiatives (tests, outreach programes)

   Exclusion criteria:

   GPs

   • Individuals who are unwilling to take part in the study.
   * Individuals with no experience in adopting new cancer tests and guidelines into practice.
   * Individuals with no experience in in detecting, managing, and referring patients with symptoms of cancer and/or are at an increased risk of developing prostate, pancreatic, GI cancer.
   * Individuals who do not adequately understand verbal explanations or written information in English.

   Patients • Individuals who are unwilling to take part in the study.

   • Individuals who do not adequately understand verbal explanations or written information in English.

   • Unable to provide written and verbal consent.

   • No direct or indirect lived experience with prostate, pancreatic, GI cancers.

   Non-clinical key stakeholders/professionals • Individuals who are unwilling to take part in the study • Individuals who are not familiar with cancer biomarkers and medical tests • Individuals with no knowledge of early detection

   • Individuals who do not adequately understand verbal explanations or written information in English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cancer detection rates | 1 year
  Whether the Man Van model can improve detection rates of prostate cancer, and reduce morbidity and mortality associated with prostate cancer, providing an economic benefit due to earlier disease detection and management.
Detection rates of other diseases | 1 year
  Whether the Man Van model can provide improved men's health services with detection of undiagnosed diabetes, blood pressure as well as lifestyle interventions (smoking, excess alcohol and weight loss advice).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D James, MBBS, FRCP, FRCR, PhD, Principal Investigator — Institute of Cancer Research/Royal Marsden NHS Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No